CLINICAL TRIAL: NCT05975541
Title: Susceptibility to Infectious Diseases in Obesity: an Endocrine, Translational, Sociological Evaluation
Brief Title: Susceptibility to Infectious Diseases in Obesity
Acronym: SIDERALE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Flavia Prodam, Associated Prof. in Clinical Nutrition and MD, Azienda Ospedaliero Universitaria Maggiore della Carita
Other Study IDs: CE277/2022
Record Dates: First submitted 2023-07-12; First posted 2023-08-04 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Obesity; Type2diabetes; Gut Microbiota; Chronic Disease
Keywords: obesity; adult; type 2 diabetes; intestinal microbiota; chronic infections; immune system
MeSH Terms: conditions — Obesity; Chronic Disease; Diabetes Mellitus, Type 2; Persistent Infection | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case (patients having chronic infections): Individuals aged between 18-65 years, presenting obesity (BMI between 30-40 kg/m2), type 2 diabetes, and chronic infections (i.e. urinary tract infections, periodontitis, herpetic infections) at the basal time.
  Interventions: Other: Observational
- control (patients without chronic infections): Individuals aged between 18-65 years, presenting obesity (BMI between 30-40 kg/m2) and type 2 diabetes.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — No intervention will be carried out in this study. Patients from both groups will be monitored for 12 months through observations at time 0, time 6 months, and 12 months. Questionnaires, good clinical practice samples, and anthropometric measurements will be made to monitor changes in the two groups.

SUMMARY:
The role of intestinal microbiota is becoming ever more important in the context of obesity, type II diabetes (T2D), and infectious disorders as represented by the emerging discipline "therapeutic microbiology". The gut microbiota is strictly interconnected with obesity and T2D playing also an important role in immune system regulation.

Obesity and diabetes can lead to chronic inflammation, which results in the secretion of pro-inflammatory cytokines like IL-6, IL-1, and TNF-alpha, causing immune system alteration which predisposes patients with obesity and T2D to chronic infections. Therefore, the principal aim of the study is to investigate changes in gut microbiota composition between patients with chronic infections or not, so as to attribute to specific phyla the formation of the infections in these patients.

DETAILED DESCRIPTION:
Obesity is nowadays a relevant public issue, with more than 650 million people affected worldwide. By definition, obesity is characterized by excessive calorie intake and lowering energy expenditure favored today by the increased sedentary lifestyle and junk food availability. Obesity represents a risk factor for cardiovascular diseases, neoplasm, and first of all type II diabetes. Nonetheless, obesity increases susceptibility to infectious disorders such as urinary tract infections, periodontitis, herpes virus infection, and also Covid-19. During the pandemic, obese patients were interested in the severe form of Covid-19 and also they presented less response to the vaccine.

Because of insulin resistance and chronic inflammation, typical of obese patients, T2D is a classical comorbidity presented by these individuals. Together these two pathologies lead to immune system deregulation and a high predisposition to secondary infections. A third player is the gut microbiota, recent discoveries demonstrated as intestinal microbiota is strictly interconnected with obesity and diabetes and with the circadian clock. Being the gut microbiota an important regulator of the immune system changes in gut microbiota composition induced by diet, obesity, and T2D can be reflected in the impairment of the immune system.

The purpose of the present study is the investigation of the gut microbiota signature in patients presenting obesity and T2D with or without infectious diseases. The idea is the identification of microbiota composition about pathological, metabolomic, and socio-economic features. Obtained results from this study could be used for the identification of new therapeutic targets involved in the development of these pathologies.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-65 years
* ability to understand the study protocol
* obesity with BMI between 30-40 kg/m2
* affects by type II diabetes
* presence/absence of chronic infections
* the possibility of equality in the two groups (matched for sex, age, and therapies)

Exclusion Criteria:

* psychological conditions that reduced the ability the comprehension of the study protocol
* subjects undergoing a diet-therapeutic regimen;
* subjects with the possibility of developing diabetic foot in the successive months
* patients with relapsing infections
* pregnancy
* bariatric surgery
* oncological and hematological pathologies
* Hypogonadism
* severe immunodepression
* vaccination in the last two weeks
* Alcohol or drug abuse
* antibiotic therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of interest for this study will be recruited by the endocrinology of the hospital "Maggiore della Carità" of Novara. The patients recruited will be equally divided into the two groups according to the presence or not of concurrent infections and will be adequately matched by age, sex, and characteristics in order to maintain a certain homogeneity of the study.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Omic signature differences between group of case and group of control | Changes in microbiota composition between time 0 months (start point of the study) and 12 months (end point of the study)
  it is expected to find differences in the signature of the gut microbiota between patients with chronic infections and those not having infections
Immune system differences between group of case and group of control | Changes in the level and type of pro-inflammatory cytokines between basal time, 0 months , 6 and 12 months (end of the study) in both case and control group
  DIfferences among pro-inflammatory cytokines (IL-6, IL-1, IL-10, IL-17, IL-18, TNF-alpha)
Patient card for the evaluation of the pharmacological therapy | changes between time 0 months (basal time) and 12 months (end of the study)
  Changes in pharmacological therapy for the treatment of diabetes, obesity, or concomitant infections due to aggravation or resolution of the pathology will be investigated through the use of a patient card.
Identification of the oral microbiota | changes in oral microbiota between the two different groups at time 0 months, 6 months and 12 months
  collection of oral microbiota by swab both in the control group and in the case
Number of white blood cells | changes in WBC biochemical levels between time 0 months, 6 months and 12 months in both case and control groups
  Use of the leucocyte formula for evaluating the number of white blood cells (WBC) in the patient's blood in both case and group.
Blood cells count | changes in blood cells count between time 0 months, 6 months and 12 months in both case and control group
  Evaluation of the blood cells with particular attention to the red blood cells in both control and case groups.
Lipid profile identification | changes in lipid profile between time 0 months, 6 months and 12 months in both case and control group
  Evaluation of the total cholesterol, LDL, and triglycerides through blood sample collection in both case and control groups.
Uric acid concentration | changes in uric acid levels between time 0 months, 6 months and 12 months in both case and control group
  Evaluation of the levels of uric acid through blood sample collection in patients.
Evaluation of urine parameters | changes in microalbuminuria and creatinuria levels between time 0 months, 6 months and 12 months in both case and control group
  Detection of the levels of microalbuminuria and creatinuria in patients of both group through urine collection and analysis.
Concentration of vitamin D | changes in vitamin D levels between time 0 months, 6 months and 12 months in both case and control group
  Detection of Vitamin D levels in patients, through blood sample collection.
Detection of immunoglobulins | changes in immunoglobulins profile between time 0 months, 6 months and 12 months in both case and control group
  Total immunoglobulins evaluation (IgE, IgA, IgD, IgG, IgM) in patients through blood sample collection. The analysis will be performed on both case and control groups.
QPE index evaluation | Changes in QPE index level between time 0 months, 6 months and 12 months in both case and control group
  Evaluation of album, alpha-1 globulin, alpha-2 globulin, beta-globulin, and gamma-globulin through protein electrophoresis (QPE) in both case and control groups.
Concentration of electrolyte levels | Changes in the electrolyte levels between time 0 months, 6 months and 12 months in both case and control group
  Detection of phosphorus and calcium levels in patients, through blood sample collection of both case and control groups.
Detection of haptoglobins level | Changes in haptoglobins levels between time 0 months, 6 months and 12 months in both case and control group
  Evaluation of the haptoglobins levels in patients through blood sample collection.
Fecal calprotectin levels identification | Changes in fecal calprotectin levels between time 0 months, 6 months and 12 months in both case and control group
  Detection of fecal calprotectin levels in stool samples collected from patients in both groups.

SECONDARY OUTCOMES:
body weight monitoring | changes between time 0 months and time 12 months
  observation of body weight differences in both case and control groups.
BMI classification | change in BMI classification between time 0 months (basal) and 12 months (end of the study)
  individuals will be obese and therefore classify based on BMI, during the study this classification could be change
evaluation of waist and hip circumference | changes between time 0 months. 6 months and 12 months
  changes in waist and hip circumference in both groups
assessment of dietary habits | changes in dietary habits between time 0 and time 12 months.
  identification of dietary habits in control groups and in the case group. Detection of the differences in the dietary habits between the two groups through the use of some specific and validated questionnaires (24h recall and Predimed).
  A 24-hour dietary recall (24HR) questionnaire to provides information about the consumption of food groups of particular interest, such as the total intake of fruits, vegetables, or added sugars.
  Predimed is a questionnaire based on adherence to the Mediterranean Diet. There is a final score that allows to identify those patients that follow this kind of nutritional regimen. Each question (if true for Mediterranean Diet) gives 1 point; the final score is structured as follows:
  ≤5 Low adherence 6 - 9= medium adherence >10 good adherence
assessment of the circadian rhythm trough MEQ questionnaire | changes in circadian rhythm between time 0 months, 6 months and 12 months
  Detection of the circadian rhythm through the Morningness Eveningness Questionnaire (MEQ) in patients of both control and case groups.
  MEQ is a self-assessment questionnaire developed to measure whether a person's circadian rhythm (biological clock) produces peak alertness in the morning, in the evening, or in between.
  The standard MEQ consists of 19 multiple-choice questions, each having four or five response options.
  Responses to the questions are combined to form a composite score that indicates the degree to which the respondent favors morning versus evening. The score is in a range between 16 and 86. If the score is lower or equal to 41 the patient is classified as an "evening" type; equal to or higher than 59, the patient is a "morning" type; between 42 and 58 is a "middle" phenotype.

CONTACTS AND LOCATIONS:
Locations (1):
- Maggiore della Carità Hospital, Novara, Italy

REFERENCES:
- See also: Related Info — https://www.who.int/data/gho/data/indicators/indicator-details/GHO/prevalence-of-obesity-among-adults-bmi-=-30-(age-standardized-estimate)-(-)
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/27356115/
- See also: Related Info — https://www.frontiersin.org/articles/10.3389/fimmu.2017.01745/full
- See also: Related Info — https://doi.org/10.1016/S0140-6736(17)32130-X
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5741209/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27388988/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22546772/
- See also: Related Info — http://eurjmedres.biomedcentral.com/articles/10.1186/s40001-020-00464-9
- See also: Related Info — https://www.frontiersin.org/articles/10.3389/fimmu.2021.621440/full
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33178196/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8624317/
- See also: Related Info — https://doi.org/10.1016/j.chom.2020.06.004
- See also: Related Info — https://www.frontiersin.org/articles/10.3389/fendo.2018.00449/full
- See also: Related Info — https://doi.org/10.1016/j.immuni.2007.01.011
- See also: Related Info — https://www.nature.com/articles/s41586-019-1171-x
- See also: Related Info — http://doi.org/10.1016/j.diabres.2020.108637
- See also: Related Info — https://www.frontiersin.org/articles/10.3389/fimmu.2020.01582/full
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9285339/?report=reader
- See also: Related Info — https://www.unboundmedicine.com/medline/citation/29492872/Intestinal_microbiota_and_the_immune_system_in_metabolic_diseases_
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32437658/
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/33298424/
- See also: Related Info — http://www.nature.com/articles/s41598-018-25168-3
- See also: Related Info — https://www.aging-us.com/article/202174/text
- See also: Related Info — http://www.frontiersin.org/articles/10.3389/fmicb.2022.939608/full
- See also: Related Info — https://genomebiology.biomedcentral.com/articles/10.1186/s13059-020-02104-1
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/31541197/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33136284/